CLINICAL TRIAL: NCT06645587
Title: Understanding and Targeting Repetitive Behaviors and Restricted Interests in Autism Spectrum Disorder Via High-Definition Transcranial Direct Current Stimulation
Brief Title: Targeting Repetitive Behaviors in Autism Spectrum Disorder Via Transcranial Direct Current Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR-2021-12375413
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; HD-tDCS; Restricted Interests; Repetitive Behaviors; Neurodevelopmental Disorders; transcranial direct current stimulation
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm Pre-SMA (Active Comparator): Active cathodal HD-tDCS over pre-SMA cortex. For HD-tDCS a 4 × 1 montage, small circular electrodes (diameter 1 cm) will be used with the cathode placed centrally over Fz with a current intensity of 0.5 mA for a total of 20 minutes (30 s ramp up/down).
  For the electrodes' placement, the investigators will follow the recommended guidelines for children.
  Interventions: Device: Active HD-tDCS over pre-SMA
- Arm left-dlPFC (Active Comparator): Active cathodal HD-tDCS over left dlPFC cortex. For HD-tDCS a 4 × 1 montage, small circular electrodes (diameter 1 cm) will be used with the cathode placed centrally over F3 with a current intensity of 0.5 mA for a total of 20 minutes (30 s ramp up/down).
  For the electrodes' placement, the investigators will follow the recommended guidelines for children.
  Interventions: Device: Active HD-tDCS over left DLPFC
- Arm Sham (Sham Comparator): Sham HD-tDCS will be delivered over pre-SMA or left-dlPFC cortex. The same electrodes placement as well as the stimulation set-up will be used as in the active stimulation conditions, but the current will be applied for 30 s and will be ramped down (0 mA) during the rest of the session without the participants awareness.
  Interventions: Device: Sham HD-tDCS

INTERVENTIONS:
Device: Active HD-tDCS over pre-SMA — Active cathodal HD-tDCS over pre-SMA cortex will be delivered for 10 days (3 sessions per week). The 4 × 1 montage using small circular electrodes (diameter 1 cm) will be applied with the cathode placed centrally over Fz. The current intensity will be set at 0.5 mA for a total of 20 minutes (30 s ramp up/down).
  Arms: Arm Pre-SMA
Device: Active HD-tDCS over left DLPFC — Active cathodal HD-tDCS over left DLPFC cortex will be delivered for 10 days (3 sessions per week). The 4 × 1 montage using small circular electrodes (diameter 1 cm) will be applied with the cathode placed centrally over F3. The current intensity will be set at 0.5 mA for a total of 20 minutes (30 s ramp up/down).
  Arms: Arm left-dlPFC
Device: Sham HD-tDCS — Sham HD-tDCS will be delivered over pre-SMA or left-dlPFC cortex for 10 days (3 sessions per week). The same electrodes placement as well as the stimulation set-up will be used as in the active stimulation conditions, but the current will be applied for 30 s and will be ramped down (0 mA) during the rest of the session without the participants awareness. Each Sham session will last 20 minutes.
  Arms: Arm Sham

SUMMARY:
Repetitive behaviors (RBs) are a prevalent feature of Autism Spectrum Disorder (ASD). There are two groups of RBs: lower-order (e.g. motor stereotypies) and higher-order RBs (e.g. restricted interests), linked to sensory-motor and the associative loops, respectively. To date, treatment options for RBs are very limited. High-definition transcranial direct current stimulation (HD-tDCS) may be effective in reducing the impact of RBs in children with ASD by targeting the associated brain alterations. Moreover, the high focality of HD-tDCS will help the investigators to disentangle the relative contribution of different brain loops (namely, sensory-motor and the associative loops) into RBs subtypes. The investigators will also study the electrophysiological patterns associated to behavioral changes after the application of HD-tDCS.

DETAILED DESCRIPTION:
The experimental design will be the following: randomized, three-arm, between subject, double blind, and placebo-controlled.

Children and adolescents with ASD will be selected and randomly assigned to three groups: 1. Active high-definition tDCS (HD-tDCS) over pre-SMA; 2. Active high-definition tDCS (HD-tDCS) left DLPFC; 3. Sham high-definition tDCS (HD-tDCS).

In this project, the investigators will work to understand whether a brain-based intervention, with the use of HD-tDCS can enhance RBs in individuals with ASD.

The protocol will allow the investigators to:

1. Test if Active high-definition tDCS (HD-tDCS) compared to sham HD-tDCS will contribute in reducing RBs
2. Test if HD-tDCS over pre-SMA cortex will decrease lower-order RBs, while HD-tDCS over dlPFC will decrease higher-order RBs
3. Test if the Active Groups will significantly improve in the remaining psychological measures compared to the Sham Group
4. Test if the Active Groups will change in the RBS-R total score will be significantly correlated with changes in neuropsychological and electroencephalographic (EEG) connectivity measures
5. Test if the Active Groups will change in the RBS-R total score will be significantly correlated with changes in the remaining psychological measures and parental stress.

The overarching goal is to provide a scientific foundation for devising new rehabilitation strategies in ASD.

ELIGIBILITY:
Inclusion Criteria:

* participants of both genders with ASD diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and based on clinical evaluation and administration of gold standard tools for ASD diagnosis
* an intelligence quotient (IQ) higher or equal to 70 (IQ ≥ 70)
* age range from 8 years to 13 years and 11 months included

Exclusion Criteria:

* the presence of neurological/medical/genetic conditions (i.e., brain tumours or genetic syndromes)
* personal or family history of epilepsy
* other primary psychiatric diagnoses (i.e., bipolar disorders, schizophrenia spectrum disorders, or adjustment disorder)
* sensorimotor deficits
* the presence of peacemaker or other metal devices in the body;
* ongoing CNS-active drug treatment
* receiving other cognitive-behavioral therapies specifically focused on RBs in the 3 months before the study

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Repetitive Behavior Scale-Revised | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The primary outcome measure will be the Total Score of the Repetitive Behavior Scale-Revised (Bodfish, 2000). It consists of a 43-item parent-report questionnaire evaluating the extent of RBs in individuals with ASD. The tool encompasses six scales: Stereotyped Behavior (6 items), Self-injurious Behavior (8 items), Compulsive Behavior (8 items), Routine Behavior (6 items), Sameness Behavior (11 items), and Restricted Behavior (4 items). The items are rated on a four-point scale (0-Behavior does not occur, 1-Behavior occurs and is a mild problem, 2-Behavior occurs and is a moderate problem, 3-Behavior occurs and is a severe problem); an overall total raw score and a total number of items score for each subscale are computed. Higher scores indicate greater severity of repetitive behaviors. The sum of all items provides a total raw score ranging from 0 to 129, with higher scores indicating more severe repetitive behaviors.

SECONDARY OUTCOMES:
Wisconsin Card Sorting Test | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The version of the Wisconsin Card Sorting Test for developmental stages evaluates executive functions. The Modified Card Sorting Test (MCST; Nelson, 1976) assesses executive functions in children aged 4-13 years. It requires assigning 48 cards, on which one to four symbols are printed in different colors and shapes. The sorting rule (number, shape, color) changes after six correct assignments. The participant must deduce the current rule from the own pattern of responses. The number of right and wrong assignments and the number of errors will be computed.
Stop Signal Task | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The Stop Signal Task is a computerized task evaluating inhibitory control. The task is structured in line with the consensus guide of SST (Verbruggen et al., 2019) and it will be performed on PsychoPy® software (Open Science Tools Ltd., Nottingham, UK). The task duration will be approximately 14 minutes. The Stop Signal Task will yield the following measures: stop signal reaction time, calculated in milliseconds by subtracting a mean Stop Signal Delays from the observed mean reaction times in no-stop trials; go accuracy; go reaction times; Stop Signal Delay.
Short Sensory Profile 2 | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The Short Sensory Profile 2 (Dunn, 2014) is a parent report questionnaire for evaluating the sensory processing pattern in children aged 3-14 years. It contains 34 items. Scores are assigned on a five-point Likert scale and range from "always = 0" to "often = 1" to "sometimes = 2" to "rarely = 3" to "never = 4". Low scores are indicative of frequent dysfunctional behavior. Based on a bell curve normed distribution, the raw score total for each quadrant can be classified as "much less than others" (lower 2%), "less than others" (between 1 SD and 2 SD below the mean, accounting for 14% of the normative sample), "just like the majority of others" (± 1 SD from the mean and accounting for 68% of the normative sample), "more than others" (between 1 SD and 2 SD above the mean), and "much more than others" (upper 2%).
Behavior Rating Inventory of Executive Function - Second Edition/ parent report | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The Behavior Rating Inventory of Executive Function (Gioia et al., 2015) is a parent report questionnaire consisting of 63 items for an ecological and comprehensive evaluation of executive functions in children aged 5-18 years. The tool encompasses 63 items evaluating inhibition, self-monitoring, shift, initiation, working memory, emotional control, planning, task-monitoring, and organization of materials. Items are further dived into 4 indices as follows: the Behavior Regulation Index, the Emotion Regulation Index, the Cognitive Regulation Index, and the Global Executive Composite. Raw scores of each scale and index are converted into T scores (M = 50, SD = 10) and percentiles. For all clinical scales and indices, T scores from 60 to 64 and from 65 to 69 are considered respectively mildly elevated and potentially clinically elevated while T scores at or above 70 are clinically significant.
Sleep Disturbance Scale for Children | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The Sleep Disturbance Scale for Children (Bruni et al., 1996) is a parent report questionnaire for evaluating the sleep functioning of children and adolescents aged 6-16 years. The tool investigates the occurrence of sleep disturbances in the previous six months throughout 26 items on a five-point Likert scale (1 = least severe and 5 = most severe). It encompasses the following scales: difficulty in initiating and maintaining sleep, sleep-disordered breathing, disorders of arousal, sleep-wake disorders, disorders of excessive somnolence, and sleep hyperhidrosis. The sum of all items provides a total raw score ranging from 26 to 130, with higher scores indicating more sleep difficulties. A T score of >70 is clinically significant while T scores under 60 or ranged 61-69 are respectively in the average or borderline range.
Child Behaviour Checklis/ 6-18 | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The Child Behaviour Checklist/ 6-18 (Achenbach and Rescorla, 2001) is a parent report questionnaire to evaluate behavioral and psychopathological symptoms during the preceding 6 months in individuals aged 6-18 years. It includes 113 items on a three-point Likert scale (0 = not true; 1 = somewhat or sometimes true; 2 = very true or often true). According to the cut-off thresholds of Achenbach and Rescorla (2001), T-scores > 69 were classified as clinically relevant, t-scores between 65 and 69 were classified as borderline, and T-scores < 65 indicated non-clinical symptoms. For the internalizing problems, externalizing problems, and total problems scales, T-scores > 63 were classified as clinically relevant, T-scores between 60 and 63 were classified as borderline, and T-scores < 60 indicated non-clinical symptoms.
Childhood Autism Rating Scale-2 | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The Childhood Autism Rating Scale-2 (Schopler et al., 2010) is a rating scale for symptoms related to ASD. Higher scores indicate more severe symptoms of ASD. The instrument is designed for children aged 2-6 years or in individuals with ASD and low functioning (IQ ≤ 79 and regardless the child's age - Standard Form), and individuals with ASD and high functioning (IQ>80 - High Functioning Form). Both versions contain 15 items rated on a 4-point scale with higher scores revealing more severe symptoms related to ASD. The total raw score is converted into standard score within three ASD severity levels: no or minimum symptoms of ASD (15-29.5 or 15-27.5 with >13 years for the standard form; 15-27.5 for the high functioning form) mild to moderate symptoms of ASD (30-30.6 or 28-34.5 with >13 years for the standard form; 28-33.5 for the high functioning form), and moderate to severe symptoms of ASD (>35 or >37 with >13 years for the standard form; >34 for the high functioning form).
Parenting Stress Index Short Form | Baseline, pre-intervention; immediately after the intervention; three-month follow-up.
  The Parenting Stress Index Short Form (Abidin, 1997) is a self-report questionnaire designed to evaluate parental stress levels in parents of children aged 1 month to 12 years. The instrument is used in both clinical and research settings. It contains 36 items rated on a five-point Likert scale (1 = strongly disagree and 5 = strongly agree). Items encompass three subscales as follows, parental distress or the experienced distress in the role of being a parent, difficult child linked to the child's behavioral problems, and parent-child dysfunctional interaction. The sum of all items results in the Total Stress score. The total raw score is converted into percentile score; percentile ≥85 is considered as clinically significant.
Electroencephalography (HD-EEG) | Baseline, pre-intervention and immediately after the intervention.
  Resting-state EEGs will be recorded in a sound-attenuated, electrically shielded room to minimize external noise and interference.

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Children Hospital, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lazzaro G, Passarini S, Battisti A, Costanzo F, Garone G, Mercier M, D'Aiello B, De Rossi P, Valeri G, Guerrera S, Casula L, Menghini D, Vicari S, Fuca E. Understanding and targeting repetitive behaviors and restricted interests in autism spectrum disorder via high-definition transcranial direct current stimulation: a study-protocol. BMC Psychiatry. 2025 Feb 25;25(1):170. doi: 10.1186/s12888-025-06506-y. PMID 40001028